CLINICAL TRIAL: NCT03954288
Title: The Serum Sclerostin Levels in Cholesteatoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ozgur Mehmet Yis, Assistant Professor Doctor, Abant Izzet Baysal University
Other Study IDs: AbantIBU-Biochem-OMY-2
Record Dates: First submitted 2019-04-30; First posted 2019-05-17 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Otitis Media Chronic; Cholesteatoma
Keywords: otitis media chronic; cholesteatoma; sclerostin
MeSH Terms: conditions — Cholesteatoma; Sclerosteosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- chronic otitis media: patients with chronic otitis media without cholesteatoma
  Interventions: Diagnostic Test: serum for sclerostin ELISA test
- cholesteatoma: patients with chronic otitis media whose cholesteatoma
  Interventions: Diagnostic Test: serum for sclerostin ELISA test
- control: patients scheduled to operation with diagnosis of other causes
  Interventions: Diagnostic Test: serum for sclerostin ELISA test

INTERVENTIONS:
Diagnostic Test: serum for sclerostin ELISA test — Blood sample to measure serum sclerostin level

SUMMARY:
The aim of this study is to investigate the levels of sclerostin in patients with cholesteatoma. So far, there is no study showing the levels of sclerostin in cholesteatoma. The investigators hope that the results of our study will start new processes that can be used in the clinic.

DETAILED DESCRIPTION:
Chronic otitis media (COM) is the perforation of the eardrum and mucosal inflammation of the space in the middle ear and the air cavities of the temporal bone over a period of three months. Although COM is defined as a multifactorial disease, its etiopathogenesis has not been fully elucidated. Cholesteatoma is a condition that disrupts the balance between bone formation and resorption in COM. The cholesteatoma is a destructive squamous epithelial lesion of temporal bone, it gradually expands and leads to serious complications by the destruction of near bone structures, ossicular chain and otic capsule. A growing debate examines the role of bone formation and destruction with osteoblasts, osteocytes and osteoclast cells in cholesteatoma formation. Sclerostin is a glycoprotein that plays a role in the regulation of bone metabolism secreted by osteocytes. Antibodies directed against sclerostin stimulate bone formation and represent a new therapeutic option for the treatment of increased bone resorption diseases, such as osteoporosis and generalized bone loss, inflammatory diseases with cartilage damage. The aim of this study is to investigate the levels of sclerostin in patients with cholesteatoma. So far, there is no study showing the levels of sclerostin in cholesteatoma. The investigators hope that the results of our study will start new processes that can be used in the clinic.

ELIGIBILITY:
Inclusion Criteria:

cholesteatoma chronic otitis media

Exclusion Criteria:

Acute infection Malignancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The experimental group of this study consisted of 75 patients who applied to AIBU Bolu Izzet Baysal Training and Research Hospital Ear Nose Throat Clinic and regularly followed up. A control group of approximately 50 people, which is demographically similar, and patients whose scheduled for operation with other causes.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
change of the levels of sclerostin in cholesteatoma at 1 month | 1 month
  So far, there is no study showing the levels of sclerostin in cholesteatoma. The investigators hope that the results of our study will initiate new processes that can be used in clinical applications.

CONTACTS AND LOCATIONS:
Locations (1):
- Özgür Mehmet Yis, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No